CLINICAL TRIAL: NCT02735759
Title: Detecting Circulating Emboli in Patients with Acute Venous Thromboembolism Using in Vivo Photoacoustic Flow Cytometry (PAFC)
Brief Title: Detecting Circulating Emboli in Patients with Acute Venous Thromboembolism
Acronym: PAFC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Required revisions were unable to be made to protocol.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 205341.
Record Dates: First submitted 2016-04-01; First posted 2016-04-13 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2018-07

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Healthy Volunteers (Other): This cohort will consist of ten healthy volunteers. The photoacoustic flow cytometry device will be used to establish device settings. The intervention with the subject will include the PAFC device to establish appropriate device settings.
  Interventions: Device: Photoacoustic flow cytometry device
- Venous Thromboembolism (Other): This cohort will consist of ten patients with newly diagnosed, non-life threatening acute venous thromboembolism. The intervention with the subjects is to perform the photoacoustic flow cytometry device to detect circulating emboli in vivo in patients with venous thromboembolism at diagnosis, during and after anticoagulation therapy.
  Interventions: Device: Photoacoustic flow cytometry device

INTERVENTIONS:
Device: Photoacoustic flow cytometry device — The device for subjects enrolled on cohort 2 will be completed on day 0 (immediately after venous thromboembolism diagnosis and prior to anticoagulation therapy), day 7 ± 3 days after initiation of anticoagulation therapy, one week ± 3 days after completion of planned anticoagulation therapy and one month ± 3 days after completion of planned anticoagulation therapy. Anticoagulation therapy is part of the patient's normal standard of care and is not part of this study however data from what therapy was received may be captured. Patients will then be followed in hematology clinic to monitor the venous thromboembolism recurrence every 3 months for one year.

SUMMARY:
The purpose of this study is to further evaluate and adjust the photoacoustic flow cytometry device and its use in detecting circulating emboli.

Study Design: Cohort 1: Normal healthy volunteers will be enrolled to further adjust the device settings. Cohort 2: Use the Phatoacoustic flow cytometry (PAFC) to detect circulating emboli in vivo in patients with venous thromboembolism at diagnosis, during and after anticoagulation therapy.

DETAILED DESCRIPTION:
Laser beam from the investigational device Phatoacoustic flow cytometry PAFC will be applied to skin and underlying blood vessels. The optical and ultrasound signal will be collected for analysis. On each tested vessel, we will estimate the vessels diameter (using optical or/and ultrasound imaging). The subject's skin pigmentation will be classified as light, medium, or dark. A photoacoustic (PA) contrast will be considered usable for detection of circulating emboli if the photoacoustic signal from the vessels is more than 1.3-fold higher than the photoacoustic signal from surrounding tissue. The device for subjects enrolled on cohort 2 will be completed on day 0 (immediately after venous thromboembolism diagnosis and prior to anticoagulation therapy), day 7 ± 3 days after initiation of anticoagulation therapy, one week ± 3 days after completion of planned anticoagulation therapy and one month ± 3 days after completion of planned anticoagulation therapy. Anticoagulation therapy is part of the patient's normal standard of care and is not part of this study however data from what therapy was received may be captured. D-dimer test will be performed on each time point as part of their normal standard of care however if the D-dimer test is not ordered as part of the standard of care it will be required for the study.. Patients will then be followed in hematology clinic to monitor the venous thromboembolism recurrence every 3 months for one year.

ELIGIBILITY:
Inclusion Criteria Cohort 1:

* Age 18 years and older
* Willing to adhere to protocol.
* Signed informed consent

Exclusion Criteria Cohort 1:

* Unable to provide informed consent.
* History of venous thromboembolism.
* Currently receiving anticoagulant therapy.

Inclusion Criteria Cohort 2:

* Ages 18 years and older
* Confirmed new diagnosis of acute venous thromboembolism.
* performance status of equal to or less than 2.
* Able to receive anticoagulation therapy.
* Willing to adhere to specific protocol requirements.
* Signed informed consent.

Exclusion Criteria Cohort 2:

* Life threatening venous thromboembolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects that posses circulating emboli. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Zhifu Xiang, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data learned from this study will be published.